CLINICAL TRIAL: NCT06851403
Title: The Effectiveness and Safety of Dupilumab in Children with Severe Asthma in China: a Real-world Study
Brief Title: The Effectiveness and Safety of Dupilumab in Children with Asthma in China: a Real-world Study
Status: Enrolling by invitation | Type: Observational
Sponsor: Guangzhou Institute of Respiratory Disease (Other)
Responsible Party: Principal Investigator, LI-HONG SUN, Guangzhou Institute of Respiratory Disease, Guangzhou Institute of Respiratory Disease
Other Study IDs: GuangzhouIRD -LSUN
Record Dates: First submitted 2024-10-03; First posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Asthma in Children
Keywords: type 2 inflammation; asthma; dupilumab
MeSH Terms: conditions — Asthma | interventions — dupilumab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Case group
  Interventions: Drug: Dupilumab

INTERVENTIONS:
Drug: Dupilumab — initial injection of 600 mg, followed by maintenance injections of 300 mg every four weeks

SUMMARY:
Observe the changes of type II inflammation markers, lung function, and symptom scores in asthmatic patients aged 6 to 14 during the use of dupilumab to analyze its efficacy.

ELIGIBILITY:
Inclusion Criteria:

Enrolled patients were required to have been on regular ICS-LABA therapy for at least 3-6 months without adequate control. The attending physician evaluated these patients as having type 2 inflammatory asthma based on factors such as FeNO (fractional exhaled nitric oxide) levels ≥ 20, sputum eosinophils (EOS) percentage ≥ 2%, and/or blood EOS count ≥ 300/μl. All children were prescribed with dupilumab during the study period.

Exclusion Criteria:

Patients with conditions other than asthma receiving treatment with dupilumab, individuals currently using other biologics or undergoing sublingual or subcutaneous immunotherapy, active parasitic infections, and children with immunodeficiency were excluded.

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The attending physician evaluated these patients as having type 2 inflammatory asthma based on factors such as FeNO (fractional exhaled nitric oxide) levels ≥ 20, sputum eosinophils (EOS) percentage ≥ 2%, and/or blood EOS count ≥ 300/μl.
Sampling Method: Probability Sample
Enrollment: 213 (Estimated)
Dates: Start 2022-01-30 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
FEV1 | From enrollment to the end of treatment through study completion, an average of 1 year
  forced expiratory volume in one second
FVC | From enrollment to the end of treatment through study completion, an average of 1 year
  forced vital capacity
FEV1/FVC | From enrollment to the end of treatment through study completion, an average of 1 year
  ratio of forced expiratory volume in onesecond to forced vital capacity
PEF | From enrollment to the end of treatment through study completion, an average of 1 year
  peak expiratory flow

SECONDARY OUTCOMES:
FeNO | From enrollment to the end of treatment through study completion, an average of 1 year
  fraction of exhaled nitric oxide
blood EOS | From enrollment to the end of treatment through study completion, an average of 1 year
  blood eosinophil count
percentage of sputum eosinophils | From enrollment to the end of treatment through study completion, an average of 1 year
TIgE | From enrollment to the end of treatment through study completion, an average of 1 year
  serum total immunoglobulin E

CONTACTS AND LOCATIONS:
Locations (1):
- Guangzhou institute of respiratory disease, Guangzhou, Guangdong, China